CLINICAL TRIAL: NCT03118206
Title: Comparison of the Effect of Lumbar Spinal Manipulation, Physical Therapy and Surgical Management in the Treatment of Lumbar Spinal Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Two authors changed their jobs.
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160804R
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Lumbar Spinal Stenosis; Spinal Manipulation; Physical Therapy; Surgery
Keywords: Lumbar spinal stenosis; spinal manipulation; physical therapy; surgery
MeSH Terms: conditions — Spinal Stenosis | interventions — Manipulation, Spinal; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lumbar spinal manipulation (Active Comparator): Lumbar spinal manipulation will be performed up to 8 times within 1 month (no more than 2 times per week) by Dr. WangTso-Liang, who is a well-trained and experienced manual therapy doctor. If the symptoms subside before the end of 1 month' treatment, the manipulation is discontinued.
  Interventions: Device: lumbar traction
- Physical therapy (Active Comparator): Physical therapy will include treatment with therapeutic exercise and modalities (lumbar traction, heattherapy, electric stimulation, and therapeutic exercise) for 2 month with frequency 3 times per week.
  Interventions: Procedure: spinal manipulation
- Surgery (Active Comparator): General anesthesia, the patient will be put in the prone and abdomen-free position. A 4-cm midline longitudinal incision will be made over the spinous processes of the L3-5 levels. It will be deepened through the fat and fascia in line with the skin incision to reach the spinous processes.The paraspinous muscles will be dissected subperiosteally down the spinous processes and along the lamina to the facet joints. Laminectomy will be done carefully at the herniated disc level for posterior decompression. The ligamentum flavum will be excised to expose the dural sac.Using blunt dissection, the investigators carefully continue down the lateral side of the dura to the floor of the spinal canal; the investigators retract the dura and its nerve root medially. After the posterior aspect of the disc space is revealed, the affected disc will be removed and discotomy will be performed.The wound will be closed in the routine fashion after meticulous hemostasis and normal saline irrigation.
  Interventions: Procedure: surgery

INTERVENTIONS:
Device: lumbar traction
  Arms: Lumbar spinal manipulation
Procedure: spinal manipulation
  Arms: Physical therapy
Procedure: surgery
  Arms: Surgery

SUMMARY:
To compare the effect of lumbar spinal manipulation, physical therapy and surgical management in the treatment of lumbar spinal stenosis.

DETAILED DESCRIPTION:
Low back pain (LBP) is a very common health problem which results in negative impact in daily life and burden especially in elderly. The global age-standardized point prevalence of LBP in 2010 was estimated to be 9.4%. Among the etiologies of low back pain, lumbar spinal stenosis is frequently encountered by physicians. In a large observational study, the prevalence of lumbar spinal stenosis was 23.6% in the general population and higher in patients more than 60 years-old. If untreated, the symptoms may persist in 70% of the patients over the 48-month observation period. On the other hand, previous studies have shown that surgery is more effective in pain relief, neurological symptoms and further functional status, however, conservative treatment still had favorable effect in patients with milder symptoms.

The role of spinal manipulation has been discussed in previous study which compared the clinical efficacy of spinal manipulation against microdiskectomy in patients with sciatica secondary to lumbar disc herniation. According to this study, the pain, disability and life quality of both groups in 12-week period had no significant difference that chiropractic spinal manipulative treatment could be considered as a primary treatment. However, comparison among the effect of spinal manipulation, physical therapy, and surgery has not been conducted before. Therefore, the purpose of this study is to compare the effect of spinal manipulation, physical therapy, and surgery in the treatment of lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 80 age years old
2. Moderate to severe low back painand/or sciatica,and/or intermittent claudication (VAS>=4)
3. Symptom duration is more than three months
4. The diagnosis is proved by MRI

Exclusion Criteria:

1. Serious spinal pathologies including spinal tumor, infection, andinflammatory disease
2. Progressive weakness, sensory loss or symptoms and signs suggesting cauda equine esion
3. Concomitant serious medical conditions
4. History of spinal surgery before
5. Severe osteoporosis or instability of the lumbar spine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
VAS pain score | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7, post-treatment 3 months and post-treatment 6 months after treatments.
  an 10-cm horizontal line will be used to assess average pain intensity in the last 1 week

SECONDARY OUTCOMES:
Modified OswestryDisability Questionnaire (MODQ) | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7, post-treatment 3 months and post-treatment 6 months after treatments.
  For evaluation of disability related to LBP, Oswestry Disability Questionnaire (ODQ) is most widely used. ODQ is a 10-item self report instrument that evaluates perceived disability in 10 areas: pain intensity, ability to lift objects, ability to walk, ability to sit, ability to stand, ability to sleep, sex life, social life, traveling, and ability to complete personal hygiene activities. By using a 6-point Likert scale (0 = no limitation; 5 = severe limitation) , the total maximum scale is doubled and reported as a percentage of the patients perceived pain-related disability, with higher scores indicating greater disability.
Swiss Spinal Stenosis Questionnaire | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7, post-treatment 3 months and post-treatment 6 months after treatments.
  The Swiss Spinal Stenosis Questionnaire is a disease-specific self-report outcome instrument commonly used in patients with lumbar spinal stenosis (LSS) for evaluation of outcomes of the treatment. It includes severity of symptoms, physical function characteristics, and patient's satisfaction after treatment. It was designed to complement existing generic measures of lumbar spine disability and health status in the evaluation of patients with LSS.
The Medical Outcome Survey Short Form (SF-36) | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7, post-treatment 3 months and post-treatment 6 months after treatments.
  The Medical Outcome Survey Short Form (SF-36) was used to assess general health status. The SF-36 measures eight dimentions of health: general health perceptions, physical function, physical role, bodily pain, social functioning, mental health, emotional role, and vitality. The eight scales may be combined into two summary scores, the physical component summary(PCS) and the mental component summary(MCS). The SF-36 has well-established psychometric properties for the general population and individuals with LBP.
Intermittent claudication | Clinical evaluation will be conducted at pre-treatment, post-treatment day 7, post-treatment 3 months and post-treatment 6 months after treatments.
  For evaluation of intermittent claudication, self-reported duration of walking will be recorded. It divides into three levels to evaluate how long the patient can walk without resting. The duration includes less than 10 minutes, 11-20 minutes, 21-30 minutes and more than 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- ShinKongHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided